CLINICAL TRIAL: NCT06621459
Title: Retrospective Observational Study of the Safety and Toxicity Management of Abemaciclib in Combination with Adjuvant Hormone Therapy in Patients with RH+ ,HER2-nonoveramplified Breast Cancer, Real-life Data
Brief Title: Retrospective Observational Study of the Safety and Toxicity Management of Abemaciclib in Combination with Adjuvant Hormone Therapy in Patients with RH+ ,HER2-nonoveramplified Breast Cancer, Real-life Data (MONARCHE29)
Acronym: MONARCHE29
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0244 - MONARCHE29
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Brest Cancer; Abemaciclib; Adjuvant Therapy; Antineoplastic Combined Chemotherapy Protocols; Breast Neoplasms
Keywords: Abemaciclib; Adjuvant Therapy; Antineoplastic Combined Chemotherapy Protocols; Breast Cancer; Real-life; Real Word Data
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Overall survival at 8 years under treatment for localized hormone-dependent breast cancer is 93.3% (1). Adjuvant therapy, especially hormone therapy, helps reduce the risk of recurrence.

However, the risk of relapse remains significant, estimated at around 20% according to studies. The SOFT study, which compares the type of hormone therapy used in premenopausal patients, estimates a relapse risk of 21.1% at 8 years (1), especially when there is initial lymph node involvement. In fact, in cases of lymph node involvement, the cumulative relapse rate at 10 years after stopping hormone therapy ranges between 19% and 36% (2), and the risk of death from breast cancer 20 years after stopping hormone therapy is estimated at 28% to 49% (2).

CDK4/6 inhibitors first demonstrated their efficacy at the metastatic stage. Abemaciclib improved median survival to 46.7 months compared to a median of 37.3 months with hormone therapy alone (Monarch 2 (3) and Monarch 3 (4)). Palbociclib showed in PALOMA-2 (5) an improvement in progression-free survival (24.8 months versus 14.5 months) without an improvement in overall survival. Ribociclib, in turn, demonstrated in MONALEESA 2 (6) an improvement in PFS (25.3 months versus 16 months) and in overall survival (63.9 months versus 51.4 months). These treatments have become the standard first-line treatment for patients with RH+ HER2 non-amplified breast cancer.

Given the results in advanced lines, CDK4/6 inhibitors have been the subject of studies in localized breast cancer, particularly in this high-risk population where the recurrence rate remains significant.

The MONARCH-E study, published on September 20, 2020 (7), led to the approval of Abemaciclib by European authorities at the time of the initial publication (median follow-up of 15.4 months) and to reimbursement starting in May 2023 after a second interim analysis (8) in this at-risk population, with a 5.6% reduction in relapse risk after 42 months of follow-up compared to hormone therapy alone.

It is crucial to clearly define the at-risk population in order to offer them treatment intensification while maintaining a satisfactory quality of life. The group benefiting from Abemaciclib presented grade III toxicity in 43% of cases and grade IV toxicity in 2.5%.

Real-world data are needed to better understand the management and toxicity of this treatment.

DETAILED DESCRIPTION:
TARGET POPULATION

Patients with high-risk RH+ HER2 non-amplified breast cancer according to the criteria of the MONARCH-E study, specifically:

Either ≥ 4 pALN (positive axillary lymph nodes)

Or 1-3 pALN and at least one of the following criteria:

* Tumor size ≥ 5 cm
* Or histological grade 3 PRIMARY OBJECTIVE

Tolerance of treatment with ABEMACICLIB in combination with hormone therapy

SECONDARY OBJECTIVES

Recurrence-free survival Safety and tolerance of treatment with ABEMACICLIB Impact of dose reduction on treatment efficacy Incidence and management of digestive toxicity Incidence of hematological toxicity Incidence of pulmonary toxicity (with radiotherapy) Tolerance data in patients over 75 years Incidence and causes of permanent discontinuation of ABEMACICLIB Quality of life data

PRIMARY EVALUATION CRITERION

Dose intensity of ABEMACICLIB treatment at 6 months SECONDARY EVALUATION CRITERIA

Median duration of ABEMACICLIB treatment Cumulative dose of treatment Frequency and severity of side effects according to CTCAE V5 classification IDFS IDFS correlated with dose reduction METHODOLOGY Multicenter retrospective study based on data

STATISTICS For the demographic analysis of the study population, quantitative variables will be represented by their mean ± standard deviation or their median ± Q1-Q3 interval depending on their distribution. Qualitative variables will be represented by the number and proportion of individuals within each category.

If necessary, quantitative variables will be compared using the Student's t-test or the Wilcoxon test depending on their distribution. Qualitative variables will be compared using the Chi-square or Fisher test depending on their distribution.

INCLUSION CRITERIA

Adult patient Patient who has received adjuvant ABEMACICLIB in combination with hormone therapy

Patient with localized RH+ HER2 non-amplified breast cancer and eligible for treatment with ABEMACICLIB according to the recommendations of the MA (Marketing Authorization) as defined below:

≥4 ipsilateral positive axillary lymph nodes OR

1 to 3 ipsilateral positive axillary lymph node(s) with at least one of the following two criteria: histological grade 3 or primary tumor size ≥5 cm

EXCLUSION CRITERIA

Patients under legal protection (guardianship, trusteeship, etc.) Refusal to participate

NUMBER OF PATIENTS Cohort consisting of all patients meeting the inclusion criteria during the study period, approximately 30 patients.

TIMELINE Inclusion duration: 23 months

Data collection period (retrospective between May 2023 and June 2025):

Study completion time (i.e., sending non-objections + data entry): 25 months

FUNDING No funding

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient who has received adjuvant ABEMACICLIB in combination with hormone therapy
* Patient with localized RH+ HER2 non-amplified breast cancer and eligible for treatment with ABEMACICLIB according to the recommendations of the MA (Marketing Authorization) as defined below:

  * 4 ipsilateral positive axillary lymph nodes OR

    1. to 3 ipsilateral positive axillary lymph node(s) with at least one of the following two criteria: histological grade 3 or primary tumor size ≥5 cm

Exclusion Criteria:

* Patients under legal protection (guardianship, trusteeship, etc.)
* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with high-risk RH+ HER2 non-amplified breast cancer according to the criteria of the MONARCH-E study, specifically:
  Either ≥ 4 pALN (positive axillary lymph nodes)
  Or 1-3 pALN and at least one of the following criteria:
  * Tumor size ≥ 5 cm
  * Or histological grade 3
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-26 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
the average dose of abemaciclib received over 6 months. | over 6 months
  The primary criterion was the average dose of abemaciclib received over 6 months.
  The average dose received was defined as: the dose administered per day, multiplied by the duration of treatment, taking into account periods of interruptions and dose reductions, divided by 183 days (6 months). This quantity can be expressed in mg/day or as a percentage of the maximum dose (full dose, without interruption).
  This criterion will be used to divide the population into two groups. The threshold of two-thirds of the maximum dose was chosen, corresponding to the reduction of the first therapeutic adjustment step. It allows separation into a group receiving a so-called full dose, corresponding to two-thirds or more of the maximum dose, and a group receiving a reduced dose, corresponding to less than two-thirds of the maximum dose. This calculation allows the identification of patients who had at least one dose adjustment

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement